CLINICAL TRIAL: NCT03794011
Title: Study to Compare 2 Minimally Invasive Fetal Neural Tube Defect Repair Techniques: Repair Using Durepair Patch vs. Repair Without Durepair Patch
Brief Title: Patch vs. No Patch Fetoscopic Meningomyelocele Repair Study
Status: Active, not recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Baylor College of Medicine (Other)
Responsible Party: Principal Investigator, Michael A Belfort, Professor and Chairman, Department of Obstetrics and Gynecology, Baylor College of Medicine
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: H-43359
Record Dates: First submitted 2019-01-02; First posted 2019-01-04 (Actual); Last update posted 2026-02-06 (Actual); Status verified 2026-02

CONDITIONS: Neural Tube Defects
Keywords: myelomeningocele; MMC; NTD; neural; defect; Spinal Bifida; Neural Tube Defect
MeSH Terms: conditions — Neural Tube Defects; Meningomyelocele | interventions — Fetoscopy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes

ARMS (1):
- fetoscopic surgical repair (Experimental): Single arm study. All patients will receive the fetoscopic repair.
  Interventions: Device: fetoscopy

INTERVENTIONS:
Device: fetoscopy — The fetoscopic arm is described above. Patients who have an appropriate window (posterior placenta) and choose fetoscopic surgery will be offered the two fetoscopic options, (i) laparotomy assisted and, (ii) totally percutaneous expandable port assisted. Patients with an anterior placenta will only be offered the lapartotomy assisted approach. All patients will undergo a fetoscopic repair of the fetal open neural tube defect including a the use of a Durepair patch.
  Other Names: Richard Wolf Medical Instruments, Corp.; Karl Storz Endoscopy-America, Inc.; Cook Medical, Inc.; Lexion Medical, LLC.; Terumo Pinnacle; Pare Surgical, Inc.; Medtronic Neurosurgery; Canon Medical; Applied Medical

SUMMARY:
The purpose of the study is to compare the maternal, fetal and neonatal outcomes of a cohort of 60 patients in whom a multilayer closure with a Durepair patch is performed with a prior cohort of patients in whom a standardized repair without patch (n = 32) was performed using the same minimally invasive fetoscopic repair technique.

The hypothesis is that there will be a thicker repair (as measured by MRI at 6 weeks post surgery) and less MMC repair dehiscence and/or CSF leak with the patch repair.

DETAILED DESCRIPTION:
Spina bifida can be a devastating neurological congenital anomaly. It results from incomplete closure of the neural tube between 22 and 28 embryological days. Its incidence is approximately 1-2 per 1,000 births. It is considered the most common congenital anomaly of the central nervous system compatible with life.

1. The most frequent form is myelomeningocele (MMC), characterized by the extrusion of the spinal cord into a sac filled with cerebrospinal fluid (CSF), and is associated with lower limb paralysis and bowel and bladder dysfunction.
2. The majority of MMCs can be diagnosed between 14 and 20 weeks of gestation. MMC is associated with Chiari II malformation, which includes a constellation of anomalies such as hindbrain herniation, brainstem abnormalities, low-lying venous sinuses and a small posterior fossa.The Chiari II malformation can have deleterious effects on motor, cranial nerve and cognitive functions. Postnatally most MMC patients develop hydrocephalus and require a ventriculoperitoneal shunt. Shunts require lifelong monitoring and have a high failure rate due to infection, obstruction, and fracture.

Experimental studies using animal models have shown that prenatal coverage of a spina bifida-like lesion can preserve neurological function and reduce or reverse hindbrain herniation.These studies suggest a "two-hit" hypothesis in which the ultimate neurologic deficit results from a combination of the failure of normal neural-tube closure (first hit) with secondary spinal cord injury resulting from prolonged exposure of sensitive neural elements to the amniotic fluid (second hit mechanism).

Based on this hypothesis, open fetal surgical repair of MMC was proposed, and the 2011 publication of the NICHD sponsored randomized controlled trial demonstrated clear neonatal benefit of open in-utero fetal surgical repair of MMC. The study showed a reduction in the incidence of hydrocephalus and in the radiographic severity of hindbrain herniation (relative risk: 0.67; 95% confidence interval: 0.56-0.81).

Open in-utero fetal surgery is not without risk and the NICHD study (MOMS Trial) showed an elevation in maternal-fetal morbidity/risk when compared to the postnatally treated group, including higher risk for chorioamniotic separation (26% vs. 0%, respectively), maternal pulmonary edema (6% vs. 0%), oligohydramnios (21% vs. 0%), placental abruption (6% vs. 0%), spontaneous membrane rupture (46%; RR: 6.15; 95% CI: 2.75-13.78), spontaneous labor (38%; RR: 2.80, 95%CI: 1.51-5.18), maternal blood transfusion (9%; RR: 7.18; 95%CI: 0.90-57.01), and preterm delivery before 34 weeks (46%; RR: 9.2; 95%CI: 3.81-22.19). The reason for the increased incidence of these complications is related to the nature of the open fetal procedure, which involves a multi-faceted invasive approach including maternal laparotomy, large hysterotomy with uterine edge stapling, and open fetal repair of the spina bifida defect that may involve manipulation and exposure of the fetus for a significant amount of time.

Fetal endoscopic surgery has progressed rapidly over the past decades and investigators are now able to perform a number of intricate procedures inside the uterus with specially designed instruments. These procedures include laser therapy for Twin-twin-transfusion syndrome, fetal cystoscopy and fulguration of posterior urethral valves, release of amniotic bands, and placement of various shunts and balloons inside fetal structures and cavities (peritoneal, pleural, cardiac, and trachea).

Fetoscopy offers a less invasive therapeutic option that could reduce a number of the morbidities (both maternal and fetal) related to open fetal procedures.

A few animal studies and growing clinical human experience with fetoscopic repair of MMC have demonstrated the feasibility of covering the defect and performing a full repair. These repairs have been accomplished using at least two (and sometimes more) entry ports through the uterine wall. Kohl et al. in Germany, have demonstrated the feasibility of performing a complete percutaneous fetoscopic repair of MMC using carbon dioxide to distend the uterus and provide a dry working area for the surgeon to perform the repair.

These investigators described a two-layer covering technique using an absorbable patch (Durasis, Cook, Germany) and sutures. However, while they showed that the procedure is feasible, their percutaneous technique with complete two layer surgical closure of the defect using sutures was associated with prolonged operative time and significant maternal and obstetrical morbidities.

Fetoscopy in a CO2 gas filled uterus has been recently reported by groups in Bonn, Germany (Kohl et al) and Sao Paulo, Brazil (Pedreira et al). The fetoscopic technique the investigators use has been developed and tested in a fetal sheep model of MMC by the investigators group and others (Peiro et al).

This fetoscopy technique has evolved over time to a 2-port technique developed by the team in Houston, Texas and its feasibility and applicability to the human uterus and fetus have been demonstrated and published (Belfort et al, 2017) and demonstrate an improved degree of flexibility in terms of access to the fetus regardless of placental location. The technique is designed to decrease the maternal risks of open uterus fetal surgery while maintaining a similar level of fetal benefit as seen in the MOMS trial.

The investigators technique employs an open abdomen/exteriorized (but closed) uterus methodology that allows the minimally invasive multi-layer closure of the fetal neural tube using the same closed skin repair currently employed at Baylor College of Medicine/Texas Children's Fetal Center using the open uterus approach. The technique employs a novel approach to low pressure uterine distention using the same carbon dioxide gas (8-12 mmHg pressure) that others attempting fetoscopic repair have used, but employing a much lower gas flow rate. In addition, the exteriorized uterus technique used by the Baylor investigators (as compared with the percutaneous method) allows improved access to the fetus in cases of anterior placentation, ability to manipulate and maintain the fetus in the required position, and optimal port placement resulting from the exteriorized maternal uterus.

In addition, because of the exteriorized uterus and the optimal placement this allows, only two access ports are needed and these can be sutured into the uterus allowing a closed seal and minimizing gas leakage. The use of humidified, warmed CO2, pioneered by the Baylor group, in fetal surgery, decreases membrane disruption and may prolong gestation without rupture of the membranes. Finally, recent advances in miniature surgical instruments (Storz 1.5 - 3mm surgical sets) allow unprecedented flexibility which enables a full surgical repair to be performed via a fetoscopic approach.

In preparation for the human trial the Barcelona group of Peiro et al tested their patch and sealant technique in a sheep model using single or double port access. Fetoscopic neural tube closure using a 12 F cannula, and when needed a second 9F cannula, a cover patch, and a medical sealant . They had similar results to that seen with open fetal surgical repair in the same sheep model.26 When they progressed to human trials this success in closing the lesion was not seen and they abandoned this approach

The team at Baylor College of Medicine/Texas Children's Fetal Center have now completed 53 cases using a 2 port exteriorized technique with results that support the initial hypothesis (Belfort et al , 2017). As with any technique there have been advances in instrumentation and technique and a multilayer closure (with or without a patch) has now been developed. The current study is designed to investigate the multilayer closure technique using a Durepair patch and to compare results to those achieved with the single layer closure.

We have recently added a percutaneous approach option for those patients with an anterior uterine window (i.e. an area of the uterine surface under the maternal anterior abdominal wall that is completely free of placenta (i.e. there is a posterior placenta or placenta that is located laterally and posterior such that the anterior uterine wall is free of placental tissue). The rationale for this is that in some selected cases, it will be possible to access the uterine surface in such a way that exactly the same port placement, membrane plication sutures and surgical repair as we currently perform, can be done through two smaller openings than the currently utilized large lower abdominal laparotomy that we use. The benefits of this proposed percutaneous approach are: Maternal - it will avoid the larger incision and reduce potential blood loss and infection risk from a long incision, reduce hospital length of stay, decrease maternal recovery and pain, and possibly give a better cosmetic outcome by avoiding a large scar. The fetal benefits will potentially include decreased heat loss from an open abdomen and thus reduced fetal hypothermia, decreased uterine artery manipulation and thus reduced risk of ischemia during the procedure, and a shortened surgery because of a much smaller length of abdominal opening to be closed.

In this protocol, All women who have an appropriate window and choose fetoscopic surgery will be offered (along with the standard open hysterotomy approach) the two fetoscopic options, (i) laparotomy assisted and, (ii) totally percutaneous expandable port assisted. In this new aspect of our protocol, the repair of the open neural tube defect will continue to follow the same principles used in open repairs currently being done at this institution and at others around the world. This involves release of the placode, dissection of the surrounding skin, development of myofascial flaps on either side of the defect, suture of the flaps over the freed placode, and attempted primary closure of the defect using available skin. The additional step in this protocol will add introduction of the Durepair patch to be laid on top of the placode prior to closure of the myofascial flaps. If necessary we will use relaxing incisions to provide additional mobility to the skin to be closed over the defect - an accepted technique routinely used in open procedures at our institution. In those cases, where we are able to complete the procedure with full skin closure of the defect, the only difference between the open uterus procedure, the laparotomy assisted fetoscopic procedure, and the totally percutaneous expandable port assisted procedure will be the approach inside the uterus. In the event of expandable port assisted repair being deemed too difficult or too risky, we will revert to laparotomy assisted fetoscopic repair, or to open repair (as has always been our alternative for any abandoned fetoscopic case).

Approximately 6 weeks after the surgery a post-procedure fetal MRI will be performed. If there is evidence of good closure of the neural tube defect and reversal of the Chiari II malformation, a vaginal delivery can be attempted based on obstetric criteria. Patients will be followed in person every 3-4 months after birth to 12 months at the Spina Bifida Clinic at TCH. Remaining visits will be yearly up to 5 years. If this is not possible, questionnaire(s) will be performed over the phone with the child's parents and records will be requested from the treating neurosurgeon on this same schedule.

ELIGIBILITY:
Inclusion Criteria:

1. Pregnant women - maternal age 18 years or older and capable of consenting for their own participation in this study.
2. Singleton pregnancy.
3. MMC with the upper boundary located between T1 and S1.
4. Evidence of hindbrain herniation (confirmed on MRI to have an Arnold-Chiari type II malformation). An exception will be made for patients unable to have an MRI due to implants or any medical reasons. These patients will have the Arnold-Chiari type II malformation reviewed by ultrasonography.
5. Absence of chromosomal abnormalities and associated anomalies
6. Gestational age at the time of the procedure will be between 19 0/7 weeks and 25 6/7 weeks.
7. Normal karyotype and/or normal chromosomal microarray (CMA) by invasive testing (amniocentesis or Chorionic Villus Sampling (CVS)). If there is a balanced translocation with normal CMA with no other anomalies the candidate can be included. Patients declining invasive testing will be excluded. Results by flouorescence in situ hybridization (FISH) will be acceptable if the patient is at 24 weeks or more.
8. The family has considered and declined the option of termination of the pregnancy at less than 24 weeks.
9. The family meets psychosocial criteria (sufficient social support, ability to understand the requirements of the study).
10. Parental/guardian permission (informed consent) for follow up of the child after birth.
11. For totally percutaneous expandable port assisted cases: Appropriate anterior window on the uterus free of placental tissue, as assessed by ultrasound, such that direct access to the fetus through the maternal abdominal wall is possible. If this criteria is not met, patient may still be eligible for laparotomy assisted fetoscopic repair if all other inclusion criteria and no exclusion criteria are met.

Exclusion Criteria:

1. Fetal anomaly unrelated to MMC.
2. Severe kyphosis.
3. Increased risk for preterm labor including short cervical length (<1.5 cm), history of incompetent cervix with or without cerclage, and previous preterm birth.
4. Placental abnormalities (previa, abruption, accreta) known at time of enrollment.
5. A pre-pregnancy body-mass index ≥40.
6. Contraindications to surgery including previous hysterotomy (whether from a previous classical cesarean, uterine anomaly such as an arcuate or bicornuate uterus, major myomectomy resection, or previous fetal surgery) in active uterine segment.
7. Technical limitations precluding fetoscopic surgery, such as uterine fibroids, fetal membrane separation, or uterine anomalies.
8. Maternal-fetal Rh alloimmunization, Kell sensitization or neonatal alloimmune thrombocytopenia affecting the current pregnancy.
9. Maternal HIV, Hepatitis-B, Hepatitis-C status positive because of the increased risk of transmission to the fetus during maternal-fetal surgery. If the patients HIV or Hepatitis status is unknown, the patient must be tested and found to have negative results before enrollment.
10. Maternal medical condition that is a contraindication to surgery or anesthesia.
11. Low amniotic fluid volume (Amniotic Fluid Index less than 6 cm) if deemed to be due to fetal anomaly, poor placental perfusion or function, or membrane rupture. Low amniotic fluid volume that responds to maternal hydration is not an exclusion criterion.
12. Patient does not have a support person (i.e. Spouse, partner, mother) available to support the patient for the duration of the pregnancy.
13. Inability to comply with the travel and follow-up requirements of the trial.
14. Participation in another intervention study that influences maternal and fetal morbidity and mortality or participation in this trial in a previous pregnancy.
15. Patient scores as severely depressed on the Edinburgh Postnatal Depression Scale
16. Maternal hypersensitivity to collagen.
17. Umbilical Cord hypercoiling or velamentous cord insertion
18. For totally percutaneous expandable port assisted cases: total anterior placentation

Ages: 18 Years to 64 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 38 (Actual)
Dates: Start 2018-12-18 (Actual); Primary Completion 2026-08 (Estimated); Study Completion 2026-08 (Estimated)

PRIMARY OUTCOMES:
MMC Repair Dehiscence and/or CSF leak | at birth
  Rate of MMC repair dehiscence and/or CSF leak in each group

CONTACTS AND LOCATIONS:
Overall Officials: Michael A. Belfort, M.D., Ph.D., Principal Investigator — Baylor College of Medicine
Locations (2):
- United States (2):
  - Stanford University: Lucille Packard's Children's Hospital, Stanford, California
  - Texas Childrens Hospital, Houston, Texas

REFERENCES:
- [Derived] Corroenne R, Mehollin-Ray AR, Johnson RM, Whitehead WE, Espinoza J, Castillo J, Castillo H, Orman G, Donepudi R, Huisman TAGM, Nassr AA, Belfort MA, Sanz Cortes M, Shamshirsaz AA. Impact of the volume of the myelomeningocele sac on imaging, prenatal neurosurgery and motor outcomes: a retrospective cohort study. Sci Rep. 2021 Jun 23;11(1):13189. doi: 10.1038/s41598-021-92739-2. PMID 34162982